CLINICAL TRIAL: NCT05729555
Title: An Open Label, Balanced, Randomized, Single-dose, Two-treatment, Two-sequence, Two-period, Two-way Crossover, Oral Comparative Pharmacokinetic (PK) Study of Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets, 400mg/50mg of Overseas Pharmaceuticals, Ltd. With Motrin IB (Ibuprofen Tablets USP 200mg (2× 200mg)) and BENADRYL (Diphenhydramine Hydrochloride Tablet 25 mg(2×25 mg)), Distributed by - Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division in Normal Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: Comparative Pharmacokinetic (PK) Study of Ibuprofen and Diphenhydramine Hydrochloride MR Tablets in Healthy Adults Under Fasting Condition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Guangzhou Kangqi Medical Technology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YYKQ-202210
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pain; Insomnia
Keywords: Ibuprofen; Diphenhydramine Hydrochloride
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders | interventions — Diphenhydramine

STUDY DESIGN:
Intervention Model Description: Test Product (T)：Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets, 400mg/50mg of Overseas Pharmaceuticals, Ltd.
  Reference Product (R)：Motrin® IB (ibuprofen tablets USP) 200mg and BENADRYL® (diphenhydramine hydrochloride tablet) 25 mg Distributed by: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets (Experimental): Specification: Each tablet containing ibuprofen 400 mg, diphenhydramine hydrochloride 50 mg Batch number: 22082801 Content: Ibuprofen 96.9%, diphenhydramine hydrochloride 102.4% Effective: August 27,2024 S torage conditions: sealed, room temperature. Manufacturers: Overseas Pharmaceuticals, Ltd. Usage and dosage：Once a day, one tablet at a time
  Interventions: Drug: reference 1 (R1): Ibuprofen Tablets (Motrin IB®)reference 2 (R2): Diphenhydramine Hydrochloride Tablets (Benadryl®)
- Motrin® IB (ibuprofen tablets USP) 200mg and BENADRYL® (diphenhydramine hydrochloride tablet) 25 mg (Active Comparator): Specification: 200 mg Batch number: 2CE2330 Content: 100.5% Expiry date: December 2023 Storage conditions; Storage in 20℃ -25℃
  Specification: 25 mg Batch number: BCC009 Content: 99.2% Effective to: December 2023 storage conditions; storage at 20℃ -25℃, shading
  Distributed by: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division Usage and dosage：Once a day, two tablets at a time
  Interventions: Drug: Compound ibuprofen polyrelease tablets

INTERVENTIONS:
Drug: Compound ibuprofen polyrelease tablets — Specification: Each tablet containing ibuprofen 400 mg, diphenhydramine hydrochloride 50 mg Batch number: 22082801 Content: Ibuprofen 96.9%, diphenhydramine hydrochloride 102.4% Effective: August 27,2024 S torage conditions: sealed, room temperature. Manufacturers: Overseas Pharmaceuticals, Ltd. Usage and dosage：Once a day, one tablet at a time
  Arms: Motrin® IB (ibuprofen tablets USP) 200mg and BENADRYL® (diphenhydramine hydrochloride tablet) 25 mg
Drug: reference 1 (R1): Ibuprofen Tablets (Motrin IB®)reference 2 (R2): Diphenhydramine Hydrochloride Tablets (Benadryl®) — Specification: 200 mg Batch number: 2CE2330 Content: 100.5% Expiry date: December 2023 Storage conditions; Storage in 20℃ -25℃ manufacturer: JOHNSON & JOHNSON CONSUMER INC. Usage and dosage：Once a day, two tablets at a time
  Specification: 25 mg Batch number: BCC009 Content: 99.2% Effective to: December 2023 storage conditions; storage at 20℃ -25℃, shading manufacturer: JOHNSON & JOHNSON CONSUMER INC Usage and dosage：Once a day, two tablets at a time
  Arms: Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets

SUMMARY:
Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets were randomized, open, two-cycle Comparative pharmacokinetic test under double crossover and fasting condition.

Main objective: Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets developed by Overseas Pharmaceuticals, Ltd.(Specification: each tablet containing ibuprofen 400 mg, Phenhenhydramine hydrochloride 50 mg) is the test preparation, JOHNSON & JOHNSON CONSUMER INC. Production (trade name: Motrin IB®, Specification: 200 mg) for comparative drug product 1, JOHNSON & JOHNSON CONSUMER INC. Hydrodramine hydrochloride (trade name: Benadryl®, Specification: 25 mg) for comparative formulation 2, In the fasting state, To investigate the pharmacokinetic parameters in healthy Chinese subjects of 1 and 2, And were compared. Secondary objective: To evaluate the safety of a single oral administration of Ibuprofen and Diphenhydramine Hydrochloride Modified-Release Tablets and reference 1 and reference 2 diphenhydramine hydrochloride tablets in fasting conditions in healthy Chinese subjects.

DETAILED DESCRIPTION:
Subjects were randomized in a 1:1 ratio to one of 2 T-R (R-T). That is, 8 subjects in the first cycle T group had fasting 1 tablet of test preparation (compound ibuprofen polyrelease tablet, specification: each containing ibuprofen 400 mg, diphenhydramine hydrochloride 50 mg, Overseas Pharmaceuticals, Ltd.; 8 subjects in the R group had fasting 1 ibuprofen tablet (200 mg) and 2 tablets of diphenhydramine hydrochloride (25 mg) with 240 ml warm water. Cross-administration after 7 days.

The 16 healthy subjects (including male and female subjects) were randomly divided into 2 groups, T-R and R-T, with 8 participants each. The selected subjects were admitted to the phase I ward of the clinical research center 1 day before each cycle and fasted for more than 10h before each cycle.

At 0 h (within 1.0 h before administration) and 5 min, 15 min, 30 min, 45 min, 1.0 h, 1.25 h, 1.5 h, 2.0 h, 2.5 h, 3.0 h, 3.5 h, 4.0 h, 4.5 h, 5.0 h, 5.5 h, 6.0 h, 7.0 h, 8.0 h, 9.0 h, 10.0 h, 12.0 h, 24.0 h, 36.0 h, and 48.0 h, Upper limb venous blood was collected at 25 time points, About 1.0 mL blood was discarded before each blood samples using intravenous indwelling needle, After each blood collection, About 4 mL of blood was collected into vacuum labeled EDTA-K2 anticoagulant.

The seated vital signs (including temperature, pulse, and blood pressure) were measured at 0 h before administration (within 1.0 h before administration) and 2.0 ± 0.5 h, 8.0 ± 0.5 h, 24.0 ± 1.0 h, 48.0 ± 1.0 h after administration. The subjects had a physical examination, vital signs, electrocardiogram and laboratory tests after the blood sampling. Medical staff during the study to observe and ask the subjects about subjective feelings and possible adverse events during the trial. If a subject has an AE during the study, the investigator should follow up the AE as far as possible until the adverse event response, or return to the screening period level, or the subject has stable condition.

ELIGIBILITY:
Inclusion Criteria:

1. The subject was fully informed of the trial purpose, nature, methods, and possible adverse effects, voluntarily acted as the subject, and signed the informed consent form prior to the start of any study procedures.
2. Healthy subjects aged 18 years or older (including 18 years old), both male and female.
3. Male weight was 50.0 kg and female weight 45.0 kg; body mass index (BMI) was within the range of 19.0 to 26.0 kg/m2 (including the cut-off value).
4. There is no birth plan and voluntary appropriate and effective contraceptive measures between the signing of the informed consent form and within 6 months after the end of the study, and no sperm donation and egg donation plan.
5. The subject was able to communicate well with the investigator and to understand and comply with the requirements of this study.

Exclusion Criteria:

1. Allergic constitution or a history of clinically significant food, drug allergy, or other allergic diseases (asthma, urticaria, eczematous dermatitis, etc.); or allergic to any component of ibuprofen or diphenhydramine; or a history of asthma or other allergic reactions after taking aspirin or other non-steroidal anti-inflammatory drugs; or allergic to ethanolamine drugs.
2. People with active upper gastrointestinal ulcer/bleeding, asthma history, or history of myasthenia gravis, angle-closure glaucoma, and prostatic hypertrophy
3. Patients with poor vascular puncture conditions, or unable to tolerate venipuncture, or a history of blood halo.
4. There are clinically meaningful diseases of cardiovascular, blood, liver, kidney, endocrine, respiratory, digestive, divine, menstrual, mental, mental, immune, skin and metabolic disorders, which are considered meaningful by the investigator, or a chronic or serious medical history of these diseases; or a surgical history that may affect the absorption and metabolism of drugs.
5. Patients with abnormal physical examination, vital signs examination, 12-lead electrocardiogram and laboratory examination, and abnormal clinical significance as judged by the study doctor.
6. human immunodeficiency virus (HIV) antibody, or hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV) antibody, or treponema pallidum antibody (anti-TP) test results are positive.
7. Women, pregnant, lactating, or women of childbearing age with unprotected sex or positive pregnancy test results within 14 days prior to planned drug administration.
8. , those who were vaccinated within 3 months before the screening (except COVID-19 vaccine), or who received COVID-19 vaccine within 1 week before the screening or who planned to receive any vaccine during the trial or 1 week after the end of the study;
9. or who donated 400 mL or received blood products or intended to donate blood (including blood components) during the trial or within 3 months after the end of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-03 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Mean residence time (MRT) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China